CLINICAL TRIAL: NCT05134727
Title: A Double-blind, Randomized, Placebo-controlled Study in Healthy Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of Oral AZD5055 Following Single and Multiple Ascending Doses
Brief Title: Assess the Safety, Tolerability and Pharmacokinetics of AZD5055 Following Single and Multiple Ascending Doses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8960C00001
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: AZD5055; Single ascending dose; Multiple ascending dose; Porcupine (PORCN) inhibitor; Healthy participants; Oral suspension
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Focal Dermal Hypoplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (single ascending doses [SAD]) (Experimental): Healthy participants will be randomized to a single dose of AZD5055 or placebo.
  Interventions: Drug: AZD5055; Drug: Placebo
- Part 2 (multiple ascending doses [MAD]) (Experimental): Healthy participants will be randomized to repeated dosing with AZD5055 or placebo
  Interventions: Drug: AZD5055; Drug: Placebo

INTERVENTIONS:
Drug: AZD5055 — Healthy participants will receive AZD5055
Drug: Placebo — Healthy participants will receive placebo

SUMMARY:
This is a phase I, First-in-Human study in healthy participants, performed at a single study center, consisting of 2 parts: Part 1 is a single ascending dose (SAD) study and Part 2 is a multiple ascending dose (MAD) study.

DETAILED DESCRIPTION:
Part 1: This is a double-blind, randomized, placebo-controlled study consisting of 2 parts. Part 1: SAD and Part 2: MAD.

Part 1 will be a double-blind, randomized, placebo-controlled study, with a sequential SAD design. Three dose levels of AZD5055 are planned to be investigated in 3 cohorts. Depending on evaluation of data from the preceding cohorts, 2 additional cohorts/dose levels may be added at the discretion of the SRC.

Part 1 will comprise of:

* A Screening Period of a maximum of 6 weeks.
* A Treatment Period during which subjects will be resident at the Clinical Unit from 1 day before IMP administration (Day 1) until at least 72 hours after IMP administration (Day 4). Subjects will receive a single oral dose of AZD5055 or placebo on Day 1.
* A Follow up Visit within 6 ± 1 day after the IMP dose.

Part 2 will be a double-blind, randomized, placebo-controlled study with a MAD design. Subjects will receive AZD5055 on Day 1 and Day 3 to Day 16, with no dosing on Day 2. Subjects will be naïve, ie, will not have participated in Part 1 of this study. Three dose levels of AZD5055 are planned to be investigated in 3 cohorts. Depending on evaluation of data of the preceding cohorts, up to 2 additional dose levels/cohorts may be added or expanded at the discretion of the SRC.

Part 2 will comprise of:

* A Screening Period of a maximum of 6 weeks.
* A treatment period with a dosing frequency (QD or BID) that will be dependent on emerging PK data from Part 1:

A) For cohorts with QD dosing regimens:

• A Treatment Period during which subjects will be resident at the Clinical Unit from 1 day before IMP administration (Day -1) until at least 72 hours after the last dose given on Day 16 (Day 19). Subjects will be dosed for a total of 15 days, receiving a single QD morning dose of AZD5055 or placebo on Day 1 and on Days 3 through Day 16.

B) For cohorts with BID dosing regimens:

* A Treatment Period during which subjects will be resident at the Clinical Unit from 1 day before IMP administration (Day -1) until at least 72 hours after the last dose given on Day 16 (Day 19). Subjects will be dosed for a total of 15 days, receiving a single morning dose of AZD5055 or placebo on Day 1 and Day 16, and repeated BID dosing on Day 3 through Day 15, 12 hours (± 30 minutes) apart.
* A Follow-up Visit within 6 ± 1 day after the last IMP dose, and an additional Follow up Visit within 29 ± 2 days after the last IMP dose.

ELIGIBILITY:
Inclusion Criteria

* Healthy male and female (of non-childbearing potential) subjects aged Part 1 (SAD): 18 - 55 years; Part 2 (MAD): 18 - 55 for male and 18 -49 for females, inclusive, with suitable veins for cannulation or repeated venipuncture.
* Female subjects must have a negative pregnancy test.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.
* Male subjects and their women of childbearing potential partners must be willing to use highly effective contraception measures and must refrain from donating sperm or fathering a child from the first day of dosing until 17 days after the last dose of Investigational medicinal product.

Exclusion Criteria

* History of any clinically important disease or disorder, or a major medical/surgical procedure or significant trauma within 4 weeks of the first dose of IMP.
* Untreated tuberculosis (TB) or a positive result for the interferon gamma release assay (ie, QuantiFERON TB Gold).
* A positive result for serum hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody, at the Screening Visit.
* Ongoing acquired or inherited immunodeficiency disorders, including but not limited to HIV or common variable immunodeficiency, or the subject is taking immune replacement therapy.
* Individuals with chronic infections (eg, urinary tract infection) or who are at increased risk of infection (eg, surgery, trauma, severe dental disease, or significant infection) within 30 days of screening.
* History of severe COVID-19 infection requiring hospitalization within the last 12 months prior to Screening, or clinical history compatible with Long COVID 19 (symptoms beyond 12 weeks of acute infection).
* Confirmed COVID-19 infection during Screening and/or admission by reverse transcription polymerase chain reaction (RT-PCR) test. Subjects who previously had a positive test result during the screening visit or on Day-1 may be reconsidered for inclusion after they recover from the infection as confirmed by a negative retest before (re-)admission.
* History of cancer within the last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed.
* History of osteoporosis, osteomalacia, Paget's disease of the bone, thyrotoxicosis, rheumatoid arthritis, Cushing's disease, or a pathological fracture.
* History of a traumatic fracture within 6 months of the Screening visit.
* A Bone density scans (DEXA scan) bone mineral density value with T-score < -1 for post-menopausal women and Z score < -1.5 for male participants and premenopausal women of non-childbearing potential subjects (MAD cohorts only).
* Has received live or live attenuated vaccine in the 30 days prior to dosing, the first dose of COVID-19 vaccine within 30 days prior to randomization, or a COVID 19 vaccine second or booster vaccination within 10 days of screening.
* Ongoing acute gastrointestinal (GI) disease, a history of chronic GI disease, ongoing acute hepatic disease, or a history of chronic hepatic disease, chronic renal disease, pancreatic disease, diabetes mellitus, or any condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of Gilbert's syndrome.
* History of muscle disease or rhabdomyolysis.
* Any laboratory values with the deviations at the Screening Visit and/or Day -1 from the reference range.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG that may interfere with the interpretation of QTc interval changes, including abnormal ST wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
* Known or suspected history of drug abuse.
* Current smokers who smoke > 5 cigarettes/e-cigarette/pipes per week or use of any tobacco in any other form.
* History of alcohol abuse or excessive intake of alcohol within 6 months prior to screening.
* Positive screen for drugs of abuse or alcohol at screening or admission.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Plasma donation within 1 month of Screening or any blood donation/loss > 500 mL within 3 months of Screening.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), HRT (for females), herbal remedies, mega dose vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Excessive intake of high caffeine-containing drinks or food (eg, coffee, tea, energy drinks).
* Has received another new chemical entity (defined as a compound that has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* Subjects who are vegans or have medical dietary restrictions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with adverse events (AEs) | Until Follow-up (7 days post dose) (approximately up to 53 days)
  To investigate the safety and tolerability of AZD5055 by assessment of AEs (non-serious and serious) following administration of SAD
Part 2: Number of participants with AEs | Until follow-up (45 days post-last dose) (approximately up to 89 days)
  To investigate the safety and tolerability of AZD5055 by assessment of AEs (non-serious and serious) following administration of MAD

SECONDARY OUTCOMES:
Part 1: Maximum observed plasma (peak) drug concentration (Cmax) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Maximum observed plasma (peak) drug concentration (Cmax) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1: profile 0-48 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Time to reach maximum observed concentration (tmax) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Time to reach maximum observed concentration (tmax) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 2: Area under plasma concentration-time curve in the dose interval (repeat dose only) (AUC[0-1τ]) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Partial area under the plasma concentration-time curve from 0 to time 12 hours post dose [AUC(0-12)] | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Partial area under the plasma concentration-time curve from 0 to time 12 hours post dose [AUC(0-12)] | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Partial area under the plasma concentration-time curve from 0 to time 24 hours post dose [AUC(0-24)] | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Partial area under the plasma concentration-time curve from 0 to time 24 hours post dose [AUC(0-24)] | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Half-life associated with terminal slope (λz) of a semi logarithmic concentration-time curve (t½λz) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Half-life associated with terminal slope (λz) of a semi logarithmic concentration-time curve (t½λz) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Mean residence time of the unchanged drug in the systemic circulation (MRTinf) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Mean residence time of the unchanged drug in the systemic circulation (MRTinf) | Day 1: profile 0-48 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Apparent volume of distribution following extravascular administration based on terminal phase (Vz/F) | Day 1: profile 0-72 hours after dose.
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Apparent volume of distribution following extravascular administration based on terminal phase (Vz/F) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Day 1-3 and Day 16-19
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Day 1-3 and Day 16-19
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Renal clearance of drug from plasma (CLR) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Renal clearance of drug from plasma (CLR) | Day 1-3 and Day 16-19
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Accumulation ratio (Rac) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Accumulation ratio (Rac) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants
Part 1: Temporal change parameter in systemic exposure (TCP) | Day 1: profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of SAD to healthy participants
Part 2: Temporal change parameter in systemic exposure (TCP) | Day 1: profile 0-48 hours after dose, Day 16; profile 0-72 hours after dose
  To characterize the PK of AZD5055 following oral administration of MAD to healthy participants

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in a sponsor approved tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8960C00001&attachmentIdentifier=fa95bc08-63d7-4b7f-8ef6-527377dab1f0&fileName=PXL_255781_Approved_CSR_synopsis_Redacted_PDF_A.pdf&versionIdentifier=